CLINICAL TRIAL: NCT03833362
Title: International, Multicenter, Randomized, Double Blind, Active-controlled, Parallel-group Phase III Study of Narlaprevir/Ritonavir and Pegylated Interferon/Ribavirin in 2 Patient Populations - naïve and Treatment Failure Patients With Genotype 1 Chronic Hepatitis C
Brief Title: Efficacy and Safety of Narlaprevir Used in Combination With Ritonavir in Treatment-Naïve and Failed Prior Treatment With Pegylated Interferon/Ribavirin Patients With Chronic Hepatitis C Genotype 1 (PIONEER - Study)
Acronym: PIONEER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: R-Pharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CJ05013008
Record Dates: First submitted 2019-02-05; First posted 2019-02-07 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — narlaprevir; Ritonavir; peginterferon alfa-2a; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NVR/RTV + PEG-INF/RBV (Treatment Naive) (Experimental): Narlaprevir - 2 tablets once a day orally
  Ritonavir - 1 capsule once a day orally
  Pegylated interferon alfa-2a/ Pegylated interferon alfa-2b - subcutaneous injection once weekly. Patients will be instructed by the investigator on how to self-administer the drug and will be given at each dispensing visit the quantity of PEG-INF alfa-2a and PEG-INF alfa-2b needed between visits.
  Ribavirin - twice daily orally. In the case of co-administration with PEG-INF alfa-2a: 5 RBV capsules (2 in the morning + 3 in the evening) or 6 RBV capsules (3 in the morning + 3 in the evening) - weight based. In the case of co-administration with PEG-INF alfa-2b: 4 RBV capsules (2 in the morning + 2 in the evening) - minimal dose or 7 (3 in the morning + 4 in the evening) - maximal dose
  Interventions: Drug: Narlaprevir; Drug: Ritonavir; Drug: Pegylated interferon alfa-2a/ Pegylated interferon alfa-2b; Drug: Ribavirin
- PEG-INF/RBV (Treatment Naive) (Active Comparator): Placebo Narlaprevir - 2 tablets once a day orally
  Placebo Ritonavir - 1 capsule once a day orally
  Pegylated interferon alfa-2a/ Pegylated interferon alfa-2b - subcutaneous injection once weekly. Patients will be instructed by the investigator on how to self-administer the drug and will be given at each dispensing visit the quantity of PEG-INF alfa-2a and PEG-INF alfa-2b needed between visits.
  Ribavirin - twice daily orally. In the case of co-administration with PEG-INF alfa-2a: 5 RBV capsules (2 in the morning + 3 in the evening) or 6 RBV capsules (3 in the morning + 3 in the evening) - weight based. In the case of co-administration with PEG-INF alfa-2b: 4 RBV capsules (2 in the morning + 2 in the evening) - minimal dose or 7 (3 in the morning + 4 in the evening) - maximal dose
  Interventions: Drug: Placebo Narlaprevir; Drug: Placebo Ritonavir; Drug: Pegylated interferon alfa-2a/ Pegylated interferon alfa-2b; Drug: Ribavirin
- NVR/RTV + PEG-INF/RBV (Treatment Failure) (Experimental): Narlaprevir - 2 tablets once a day orally
  Ritonavir - 1 capsule once a day orally
  Pegylated interferon alfa-2a/ Pegylated interferon alfa-2b - subcutaneous injection once weekly. Patients will be instructed by the investigator on how to self-administer the drug and will be given at each dispensing visit the quantity of PEG-INF alfa-2a and PEG-INF alfa-2b needed between visits.
  Ribavirin - twice daily orally. In the case of co-administration with PEG-INF alfa-2a: 5 RBV capsules (2 in the morning + 3 in the evening) or 6 RBV capsules (3 in the morning + 3 in the evening) - weight based. In the case of co-administration with PEG-INF alfa-2b: 4 RBV capsules (2 in the morning + 2 in the evening) - minimal dose or 7 (3 in the morning + 4 in the evening) - maximal dose
  Interventions: Drug: Narlaprevir; Drug: Ritonavir; Drug: Pegylated interferon alfa-2a/ Pegylated interferon alfa-2b; Drug: Ribavirin
- PEG-INF/RBV (Treatment Failure) (Active Comparator): Placebo Narlaprevir - 2 tablets once a day orally
  Placebo Ritonavir - 1 capsule once a day orally
  Pegylated interferon alfa-2a/ Pegylated interferon alfa-2b - subcutaneous injection once weekly. Patients will be instructed by the investigator on how to self-administer the drug and will be given at each dispensing visit the quantity of PEG-INF alfa-2a and PEG-INF alfa-2b needed between visits.
  Ribavirin - twice daily orally. In the case of co-administration with PEG alfa-2a: 5 RBV capsules (2 in the morning + 3 in the evening) or 6 RBV capsules (3 in the morning + 3 in the evening) - weight based. In the case of co-administration with PEG alfa-2b: 4 RBV capsules (2 in the morning + 2 in the evening) - minimal dose or 7 (3 in the morning + 4 in the evening) - maximal dose
  Interventions: Drug: Placebo Narlaprevir; Drug: Placebo Ritonavir; Drug: Pegylated interferon alfa-2a/ Pegylated interferon alfa-2b; Drug: Ribavirin

INTERVENTIONS:
Drug: Narlaprevir — yellow film-coated 100 mg. tablets
  Arms: NVR/RTV + PEG-INF/RBV (Treatment Failure); NVR/RTV + PEG-INF/RBV (Treatment Naive)
Drug: Ritonavir — 100 mg tablets encapsulates in gelatin capsules (for blinding purposes)
  Other Names: Norvir
  Arms: NVR/RTV + PEG-INF/RBV (Treatment Failure); NVR/RTV + PEG-INF/RBV (Treatment Naive)
Drug: Placebo Narlaprevir — yellow film-coated 100 mg. tablets identical to Narlaprevir tablets
  Arms: PEG-INF/RBV (Treatment Failure); PEG-INF/RBV (Treatment Naive)
Drug: Placebo Ritonavir — 100 mg lactose/ cellulose tablets encapsulated in gelatin capsules (for blinding purposes) identical to Ritonavir capsules
  Arms: PEG-INF/RBV (Treatment Failure); PEG-INF/RBV (Treatment Naive)
Drug: Pegylated interferon alfa-2a/ Pegylated interferon alfa-2b — 180µg for subcutaneous injections in 0.5 ml syrettes / 1.5 µg/kg for subcutaneous injections in 50µkg, 80µkg,100µkg, 120µkg, 150µkg in vials
  Other Names: Pegasys; PegIntron
Drug: Ribavirin — hard gelatin, white 200mg. capsules
  Weight-based dose was 1000 mg/day (patient weight <75 kg) or 1200 mg/day (patient weight ≥75 kg) with Peginterferon alfa-2a and 800 mg/day (patient weight <65 kg) - 1400 (patient weight >105 kg) mg/day with Peginterferon alfa-2b
  Other Names: Rebetol

SUMMARY:
The purpose of this study was to confirm that combination of narlaprevir (NVR) and ritonavir (RTV) used as a metabolic inhibitor with pegylated interferon (PEG-INF) and ribavirin (RBV) leads to a superior Sustained Virological Response (SVR) rate compared to treatment with pegylated interferon and ribavirin in treatment-naïve and treatment failure patient populations.

DETAILED DESCRIPTION:
The study included 3 time periods:

* Screening period with duration up to 3 weeks during which study eligibility was confirmed.
* Double-blind treatment period: all eligible patients divided into Treatment naive and Previous treatment failure subpopulations were randomized in one of the two parallel treatment arms in 2:1 ratio:

  1. Arm 1: All patients received the combination of NVR/RTV + PEG-INF/RBV for 12 weeks that was followed by PEG-INF and RBV for 12 weeks (total treatment duration of 24 weeks).
  2. Arm 2: Therapy with PEG-INF and RBV (standard of care) for 48 weeks with placebo equivalent for NVR and RTV for the first 12 weeks.

     Different types of pegylated interferon could be used for treatment. The assignment to the pegylated interferon alfa-2a or pegylated interferon alfa-2b treatment will be also performed using web system, in a 1:1 ratio.

     Clinical efficacy of each arm were assessed 24 weeks after the end of treatment with undetectable hepatitis C virus (HCV) RNA by lower limit of detection (LOD) 24 weeks following the end of treatment. In case of serum HCV-RNA levels were greater than or equal to 100 IU/mL at Week 12 of treatment (Arm 1) or serum HCV RNA declined from baseline less than 2 log after 12 weeks of treatment or serum HCV-RNA levels ≥LOD at week 24 of treatment (Arm 2) patients were considered non-responders and discontinued participation in the study. In case of satisfactory treatment response all patients were additionally administered with PEG-INF/RBV for 12 weeks (total of 24 weeks of treatment) in Arm 1, and for 36 weeks (total of 48 weeks of treatment) in Arm 2.
* Follow-up period during which patients do not receive any study medication. The duration of the follow-up period after the end of study treatment will be 24 weeks.

Overall, each patient will participate in the study for approximately up to 75 weeks from the time the patient signs the Informed Consent Form through the final visit

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≥ 40 and ≤ 125 kg;
* Documented infection with HCV genotype 1 (Mixed infections with other genotypes are not eligible):

  1. treatment naïve (to interferon and ribavirin); or
  2. treatment failure patients (patients must have received interferon/ribavirin at standard doses for a minimum of 12 weeks);
* Minimum HCV-RNA level of ≥10,000 IU at baseline;
* No evidence of cirrhosis; availability at Baseline of at least one of the following tests negative results:

  1. Liver biopsy showing no cirrhosis (not later than within 3 years prior to Baseline) or
  2. FibroScan elasticity score < 12.5 kPa 12 months prior to baseline or
  3. FibroTest < 0.75 12 months prior to baseline and aspartate aminotransferase (AST)/platelet ratio (APRI) of ≤ 1 during screening
* Using acceptable contraception methods for both partners from enrollment into the study until 6 months following the end of treatment;
* Willingness to give written informed consent.

Exclusion Criteria:

* Previous treatment with any HCV NS3-specific protease inhibitor and/ or other direct antiviral agents (e.g. HCV polymerase inhibitors);
* Treatment for HCV infection 30 days before the enrolment;
* Use of prohibited medications within 2 weeks prior to start of study medications (inducers or substrates of CYP3A4);
* Findings suspicious for hepatocellular carcinoma (HCC);
* Hepatic failure at present or in history;
* Auto-immune hepatitis in history;
* Anti-nuclear antibodies (ANA) titers > 1:320;
* Evidence of gallstones, choledocholithiasis and calcified gallbladder;
* HBsAg positive;
* HIV positive;
* Serum hemoglobin of <13g/dL for males and <12g/dL for females;
* Neutrophils <1500/mm3 (<1,5х109/L) at Screening;
* Platelets <150000/mm3 (<150х109/L) at Screening (patients with a platelet count >100,000/mm3 (>100х109/L) but less than 150,000/mm3 (150х109/L) can be included in the study in case a Fibroscan or FibroTest or liver biopsy during the study screening period shows no cirrhosis)
* Total bilirubin >1.6 mg/dL (>27.36 µmol/L) unless history of Gilbert's disease. If Gilbert's disease is the proposed etiology, this must be documented in the subject's chart;
* Direct bilirubin >1.5 x upper limit of normal (ULN) of the laboratory reference range at Screening;
* Serum albumin < lower limit of normal (LLN) of laboratory reference range at Screening;
* Serum creatinine >ULN of the laboratory reference at Screening;
* Serum aspartate aminotransferase (AST) / alanine aminotransferase (ALT) >5 x ULN of the laboratory reference range at Screening;
* Thyroid stimulating hormone (TSH) >1.2 ULN or <0.8 LLN;
* Contraindications to pegylated interferon, ribavirin and/or ritonavir treatment;
* Hypersensitivity to any of the study drugs;
* Active or suspected cancer;
* Psychiatric disease (moderate or severe depression, schizophrenia, bipolar disorder et al);
* Previous suicide attempt or suicidal ideation;
* Drug addiction;
* Opiate agonist substitution therapy;
* History of active gout within the past year;
* Organ transplant (except of cornea and hair transplant);
* Pregnant or nursing women;
* Men whose female partners are pregnant or planning pregnancy;
* Any medical condition that could interfere with the patient's participation and completion of the study;
* Use of other investigational drugs/ participation in other clinical trial within 30 days before the enrolment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2014-05-07 (Actual); Primary Completion 2016-03-23 (Actual); Study Completion 2017-02-21 (Actual)

PRIMARY OUTCOMES:
Number of patients with Sustained Virologic Response (SVR24) | Week 24 after the end of treatment
  HCV RNA undetectable by Limit of detection (LOD)

SECONDARY OUTCOMES:
Number of patients who achieve the Rapid Virological Response (RVR) | Week 4 of treatment
  HCV RNA < LOD
Number of patients who achieve the Early Virological Response (EVR) | Week 12 of treatment
  HCV RNA <LOD
Number of patients who achieve the End of Treatment Response (ETR) | Week 24 of treatment (Arm 1), Week 48 of treatment (Arm 2)
  HCV RNA <LOD
Number of patients who achieve the SVR12 | Week 12 after the end of treatment
  HCV RNA undetectable (by LOD)
Number of patients who develop viral breakthrough | Week 24 of treatment (Arm 1), Week 48 of treatment (Arm 2)
  Greater than or equal to 1 log10 increase in HCV-RNA above nadir, or detectable HCV-RNA, while on treatment after an initial drop below detection
Number of patients who develop relapse | Week 24 after the end of treatment
  HCV RNA undetectable by LOD at end of treatment with subsequent detectable HCV RNA
Number of patients who develop anemia | Week 24 of treatment (Arm 1), Week 48 of treatment (Arm 2)
  Anemia is defined as as Hb <10g/dL
Number of patients who develop neutropenia | Week 24 of treatment (Arm 1), Week 48 of treatment (Arm 2)
  Neutropenia is defined as neutrophils <0.75x109/L

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — R-Pharm
Locations (20):
- Russia (20):
  - South-Ural State Medical University, Clinic of Medical Academy, Infectious Diseases Department, Chelyabinsk
  - Kazan State Medical Academy, Republican Clinical Hospital of Infectious Diseases n.a. A.F. Agafonov, Kazan'
  - Federal Budget Science Institution Central Science and Research Institute of Epidemiology of RosPotrebNadzor, Moscow
  - Federal State Budget Healthcare Institution Central Clinical Hospital of Russian Academy of Science, Moscow
  - First Moscow State Medical University n.a. I.M. Sechenov, Clinic of Nephrology, Internal and Professional Diseases n.a. E.M. Tarleev, Moscow
  - First Moscow State Medical University n.a. I.M. Sechenov, Propedeutics of Internal Diseases Department, Moscow
  - Moscow State Medical Stomatological University n.a. A. I. Evdokimov, Clinical Infectious Hospital #1, Clinical Infections Department, Moscow
  - Public Corporation "Clinical Hospital of Centrosouze", Moscow
  - Public Corporation "MedElitConsulting", Moscow
  - State Budget Healthcare Moscow Institution Clinical Scientific Center of Healthcare Department of Moscow, Moscow
  - State Budgetary Healthcare Organization Clinical city hospital #24, Moscow
  - Novosibirsk State Medical University, Clinical city hospital #12, Therapeutic Department, Novosibirsk
  - Military Medical Academy of Ministry of Defense of Russian Federation n.a. S.M. Kirov, Infectious Diseases Department, Saint Petersburg
  - Saint Petersburg State Budget Healthcare Institution Center of AIDS and Infectious Diseases Prevention and Control, Saint Petersburg
  - Saint Petersburg State Budgetary Healthcare Institution Clinical Hospital of Infectious Diseases n.a. S.P. Botkin, Saint Petersburg
  - Clinic of Samara State Medical University, Department of Infectious Diseases, Samara
  - Public corporation Medical company "Gepatolog", Samara
  - Municipal Healthcare Institution Clinical city hospital #2 n.a. V.I. Razumovsky, Infectious Diseases Department, Saratov
  - Stavropolsky Krai Clinical Hospital, Gastroenterology Department related to Hospital Therapy Department, Stavropol
  - Stavropolsky State Medical University, Clinic of Gastroenterology, Hepatology and Pancreatology, Stavropol